CLINICAL TRIAL: NCT03110250
Title: A Nation-wide Registry of Familial Hypercholesterolemia : Clinical Status in Turkey (A-HIT2)
Brief Title: Familial Hypercholesterolemia in Turkey (A-HIT2)
Acronym: A-HIT2
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Collaborators: Turkish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Meral Kayikcioglu, Professor MD, Ege University
Other Study IDs: A-HIT2
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Familial Hypercholesterolemia; Atherosclerosis
Keywords: Familial Hypercholesterolemia; registry; Turkey; Lipid lowering therapy
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A-HIT2, is also designed as a National FH registry. At least 1000 FH patients will be recruited from 30 outpatient clinics representing the 12 Nuts statistical Regions in Turkey proportional to the 2015 Turkey's Population distribution.[14] Both HeFH and HoFH patients are eligible for enrollment. Sites specialized on cardiology, internal medicine, and endocrinology were invited by the Turkish Society of Cardiology.

DETAILED DESCRIPTION:
At least 1000 FH patients will be recruited from 30 outpatient clinics representing the 12 Nuts statistical Regions in Turkey proportional to the 2015 Turkey's Population distribution. Both HeFH and HoFH patients are eligible for enrollment. Sites specialized on cardiology, internal medicine, and endocrinology were invited by the Turkish Society of Cardiology. The primary objective of this cross-sectional study, is to detect the clinical status and management of the patients diagnosed with FH in Turkey. The secondary objectives are; to detect the pattern of clinical presentation, to know the medication use, to define the clinical response to LLT, to evaluate the attainment of LDL-cholesterol goals and to identify resistance and/or intolerance to LLT. Defining the CV risk factors and approach to these factors by the physicians, and comparing the attitudes in different specialty groups (cardiology, endocrinology and internal medicine) are also among the secondary objectives of the registry. Eligibility for screening was defined as having LDL-cholesterol levels > 160 mg/dl either as on treatment or untreated values. Centers may enroll both incident and prevalent patients. The inclusion criteria included age > 18 years and being diagnosed as possible FH. The possible FH was defined as having a total score of > 2 according to Dutch lipid clinic network (DLCN) criteria. Patients with triglyceride levels > 400 mg/dl or secondary hyperlipidemia (ie, untreated hypothyroidism, nephrotic syndrome, cholestasis, etc..) will be excluded from the study. Two different data sets will be collected for A-HIT2. The physicians will complete electronic case report forms for each patient Patients will also complete a short survey to assess the level of disease awareness. This survey is also designed to give information on the patients' perceptions and knowledge on cholesterol, its harm, and LLT. All data will be collected in a single visit. Data verification will be based on the source document control of 5% sample randomly selected per center.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years and being diagnosed as possible FH.
* The possible FH was defined as having a total score of > 2 according to Dutch lipid clinic network (DLCN) criteria

Exclusion Criteria:

* Patients with triglyceride levels > 400 mg/dl or secondary hyperlipidemia (ie, untreated hypothyroidism, nephrotic syndrome, cholestasis, etc..) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 1000 Familial Hypercholesterolemia (FH) patients are being recruited from 30 outpatient clinics representing the 12 Nuts statistical Regions in Turkey proportional to the 2015 Turkey's Population distribution. Both HeFH and HoFH patients are eligible for enrollment. Sites specialized on cardiology, internal medicine, and endocrinology were invited by the Turkish Society of Cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-02-26 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
number of patients receiving proper treatment for FH | February- November 2017
  how many patients are receieving the proper lipid lowering drugs for the diagnosis of FH

SECONDARY OUTCOMES:
number of patients reaching LDL-cholesterol goal according to risk status (risk level) | February- November 2017
  how patients diagnosed with FH in Turkey are managed, that is to what percent they reach ldl goals.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Kayikcioglu, Principal Investigator — Ege University
Locations (1):
- Ege University Medical School, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No